CLINICAL TRIAL: NCT00767104
Title: A Study to Evaluate the Efficacy of Silk - Like Bedding Fabric, as Used in a Standard Pillow Case, in the Treatment of Acne Vulgaris
Brief Title: Efficacy of Silk - Like Bedding Fabric Pillow Case in the Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Precision Fabrics Group, Inc. (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00006471; 33685 (Other: WakeForest)
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silk-Like Pillowcase (Experimental): Silk- Like pillowcase-One-half of subjects will be assigned to sleep on the study product, which is a standard size pillowcase made of a silk-like fabric every night for 12 weeks. The study pillowcases are fabricated from a light-weight plain-weave fabric woven of 100 percent synthetic yarns. The fabric is comprised of approximately 50% polyester and 50% nylon. The yarns in the fabric are formed from continuous-filament fibers, with no fibers projecting beyond the planar surface of the fabric. The antimicrobial technology used in the fabric is incorporated into the fibers during the finishing process and does not migrate out of the fabric or cause adverse reactions with skin contact.
  Interventions: Other: Silk like Pillowcase
- Cotton Pillowcase (Placebo Comparator): Placebo Comparator-One-half of subjects will be assigned to sleep on the placebo pillow case every night for 12 weeks. Placebo pillowcase is made of 100% cotton
  Interventions: Other: Cotton Pillowcase

INTERVENTIONS:
Other: Silk like Pillowcase — sleep on silk-like pillowcase each night
  Arms: Silk-Like Pillowcase
Other: Cotton Pillowcase — Sleep on placebo cotton pillowcase each night
  Arms: Cotton Pillowcase

SUMMARY:
The purpose of this research study is to better understand how this study pillowcase works when people use it to treat acne. Most people, including people with acne, sleep six to eight hours each night in direct contact with bedding fabrics that provide no benefit to the healing process associated with acne. The fabric in this study pillowcase may be able to reduce bacteria on the skin. This study would evaluate how acne is affected by this silk-like pillowcase. This type of study has not been done before.

DETAILED DESCRIPTION:
This is a pilot study of subjects with mild to moderate/severe facial acne vulgaris with an assessment of 2-4 on the Investigator Global Assessment (IGA) scale . We will enroll 40-60 subjects in order to obtain 40 evaluable subjects. Evaluable subjects will be defined as those that complete the protocol, or those that fail to complete due to an adverse event related to the study. One-half of subjects will be assigned to sleep on the study product, which is a standard size pillowcase made of a silk-like fabric. The other half will be assigned to sleep on the placebo pillowcase made of 100% cotton. Each subject will be instructed to sleep on this pillowcase every night for 12 weeks. Investigators will be blinded to the type of pillowcase used by the study subject. The distribution of placebo and study product pillowcases will be randomized 1:1. The study period will last for 12 weeks. Subjects will be evaluated at baseline, weeks 2, 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with facial acne vulgaris, 12 years of age or older, that agree to participate and provide written consent
* Greater than 5 superficial inflammatory lesions with less than 3 nodules on the face
* A score of 2-4 on the Investigator Global Assessment
* Women of childbearing potential will be allowed to participate in the study, and these subjects will be required to use at least one form of birth control
* Female subjects will have a urine pregnancy test if applicable.

Exclusion Criteria:

* Use within 4 weeks of baseline of systemic anti-inflammatory medication, which may influence study outcome, such as systemic corticosteroids
* Application or use within 2 weeks of baseline of topical acne or rosacea medications or topical anti-inflammatory medication, which may influence study outcome
* Presence of a concurrent medical condition, which is determined by the investigator to potentially interfere with study outcomes or patient assessments
* Subjects who have taken isotretinoin within the past 6 months
* Subjects with known allergy or sensitivity to polyester or nylon fibers in fabric
* Pregnant women and women who are breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan B Fleischer, MD, Principal Investigator — Wake Forest University Health Sciences, Dermatology

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for this study from 10/01/08 through 11/25/08. Cable TV advertising was the route of recruiting subjects and our patient database at Wake Forest University Dermatology Clinical Studies.
Groups:
- DermaTherapy Pillowcases: The study pillowcases are fabricated from a light-weight plain-weave fabric woven of 100 percent synthetic yarns. The fabric is comprised of approximately 50% polyester and 50% nylon. The yarns in the fabric are formed from continuous-filament fibers, with no fibers projecting beyond the planar surface of the fabric. The antimicrobial technology used in the fabric is incorporated into the fibers during the finishing process and does not migrate out of the fabric or cause adverse reactions with skin contact.
- Control Pillowcase: placebo pillowcase made of 100% cotton
Period: Overall Study
Arm/Group | DermaTherapy Pillowcases | Control Pillowcase
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DermaTherapy Pillowcases | Control Pillowcase | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Total Lesion Count
Description: The number of papules, pustules and cysts at Week 12.
Time Frame: 12 weeks
Population: Number of participants in each group
Measure: Mean (95% Confidence Interval); unit: lesions
Groups:
- Experimental Silk-like Pillowcases: The study pillowcases are fabricated from a light-weight plain-weave fabric woven of 100 percent synthetic yarns. The fabric is comprised of approximately 50% polyester and 50% nylon. The yarns in the fabric are formed from continuous-filament fibers, with no fibers projecting beyond the planar surface of the fabric. The antimicrobial technology used in the fabric is incorporated into the fibers during the finishing process and does not migrate out of the fabric or cause adverse reactions with skin contact.
- Control Cotton Pillowcase: placebo pillowcase made of 100% cotton
Arm/Group | Experimental Silk-like Pillowcases | Control Cotton Pillowcase
Number analyzed (Participants) | 20 | 20
lesions | 36.6 [22.9 to 50.3] | 30.7 [18.7 to 42.6]

2. Secondary Outcome: % Reduction in Total Lesion Count
Description: .This is a measure of the % reduction in the total number of papules, pustules and cysts at Week 12.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: % reduction in total lesion count
Arm/Group | DermaTherapy Pillowcases | Control Pillowcase
Number analyzed (Participants) | 20 | 20
% reduction in total lesion count | 13.1 [2.3 to 23.9] | 21.7 [12.5 to 31.0]

ADVERSE EVENTS:
Arm/Group | DermaTherapy Pillowcases | Control Pillowcase
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Results limited by low number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No